CLINICAL TRIAL: NCT06472349
Title: Structure and Function of the Upper Trapezius and Its Role in Chronic Shoulder Pain: an Investigation of Kinematics, Morphology, Muscle Quality and Activation Distribution
Status: Recruiting | Type: Observational
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, National Yang Ming Chiao Tung University
Other Study IDs: NYCU112175AE
Record Dates: First submitted 2024-06-02; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Chronic Shoulder Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic shoulder pain group
- Healthy control group

SUMMARY:
Prior research has explored factors influencing muscle activation, including muscle thickness, fear avoidance beliefs (kinesiophobia), and somatosensory integration. In individuals with chronic shoulder pain, various characteristics impacting symptoms and treatment outcomes have been identified, such as psychosocial factors, fear avoidance, central sensitization, somatosensory impairments, and brain morphology changes. These shared characteristics affecting both muscle activation and chronic shoulder pain may potentially modulate upper trapezius muscle activation during functional movements in patients with chronic shoulder pain. Notably, there remains a gap in the literature concerning investigations into the upper trapezius muscle's morphology and quality, fear avoidance, central sensitization, somatosensory impairments, and their interplay with upper trapezius muscle activation in chronic shoulder pain patients.

To address these gaps, this study aims to: this study aims to: 1) compare different methods of measuring clavicular kinematics using an electromagnetic tracking system; 2) establish the reliability and validity of measuring muscle thickness and fat infiltration through ultrasound and magnetic resonance imaging; 3) compare shoulder kinematics, muscle activation, muscle morphology, and muscle fat infiltration in individuals with chronic shoulder pain with matched healthy controls; 4) explore the correlation between the factors that may influence upper trapezius muscle activation, including basic data of the subjects, muscle morphology, and muscle fat infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Chronic shoulder pain group

  * 18-50 years old18-50 years old
  * unilateral and non-traumatic shoulder pain
  * pain duration longer than 3 months
  * pain intensity more than VAS=2 during movement
  * presence 3 of 5 positive pain provocation tests: Hawkins-Kennedy test, Jobe test, or Neer's test Painful Arc, and Resistance Test against External Rotation.
* Healthy control group

  * presenting no shoulder pain at rest or during daily activities
  * negative results of the pain provocation test: Hawkins-Kennedy test, Jobe test, Neer's test, Painful Arc, Resistance Test against External Rotation and Spurling's neck compression test.

Exclusion Criteria:

- Chronic shoulder pain group

* history of significant shoulder trauma, such as fracture or ultrasonography clinically suspected full thickness cuff tear
* recent shoulder dislocation in the last 2 years
* diagnosis of adhesive capsulitis characterized by a gradual and painful loss of both active and passive ROM in all shoulder planes, primarily external rotation
* shoulder pain originating from the cervical spine by using Spurling's neck compression test
* shoulder pain owing to the following disorders: arthritis (e.g., rheumatoid arthritis, osteoarthritis of shoulder complex), neurologic (e.g., stroke), neoplastic (e.g., breast cancer). and/or referred pain (e.g., visceral referred pain)
* corticoid injections over the shoulder during 6 months prior to the study
* history of shoulder and neck surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Shoulder kinematics | During the procedure
  The scapular kinematics will be assessed, including scapular internal/external rotation, upward/downward rotation, and posterior/anterior tilt angle. Clavicular kinematics will be evaluated by measuring clavicular protraction/retraction, elevation/depression, and posterior rotation angle.
Muscle activation | During the procedure
  The average root mean square (RMS) value collected from surface EMG and outcomes collected by high-density EMG including average root mean square (RMS) value in whole/upper/lower regions, the RMS value distribution, and position of the barycentre of RMS distribution in different humeral elevation angles and different isometric shoulder and scapular tasks will be the outcome measures related to muscle activation.

SECONDARY OUTCOMES:
Oscillation frequency | During the procedure
  The oscillation frequency (Hz) of the muscle obtained from the myotonometer will represent the muscle tone
Dynamic stiffness | During the procedure
  The dynamic stiffness (N/m) of the muscle obtained from the myotonometer will represent the muscle tone
Mechanical stress relaxation time (ms) | During the procedure
  The mechanical stress relaxation time (ms) of the muscle obtained from the myotonometer will represent the muscle tone
Muscle thickness and cross-sectional area | During the procedure
  The upper, middle and lower trapezius muscle thickness and cross-sectional area obtained from MRI and the upper, middle and lower trapezius muscle thickness obtained from musculoskeletal sonography.
Muscle thickness change at rest and in contraction | During the procedure
  The muscle thickness at rest, during arm raise at 90o abduction, during 2-kg abduction, during 4-kg abduction, and the change (%) between the latter three and at rest.
Muscle fat quantification | During the procedure
  The upper, middle and lower trapezius muscle fat quantification indicate the muscle fat infiltration.
Muscle / fat fraction | During the procedure
  The upper, middle and lower trapezius muscle / fat fraction indicate the muscle fat infiltration.
Echo intensity | During the procedure
  The echo intensity of the upper, middle and lower trapezius muscle obtained from the musculoskeletal sonography.
Pain intensity | During the procedure
  The score obtained from the VAS scale and NRPS scale during the most painful movement represent the pain intensity of the chronic shoulder pain group.
Disability level | During the procedure
  The FLEX-SF score and DASH score will indicate the disability level of the subjects.
Craniovertebral angle | During the procedure
  The cranial-vertebral angle will indicate the level of forward head posture.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan